CLINICAL TRIAL: NCT02988050
Title: Propofol-dexmedetomidine Versus Propofol-remifentanil Conscious Sedation for Awake Craniotomy During Epilepsy Surgery
Brief Title: Conscious Sedation for Epilepsy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Dr Ezzeldin Ibrahim, Assistant Professor in anaesthesia, intensive care, and pain medicine, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MenoufiaU2016
Record Dates: First submitted 2016-11-28; First posted 2016-12-09 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Epilepsy
Keywords: Epilepsy Surgery; Conscious sedation
MeSH Terms: conditions — Epilepsy | interventions — Remifentanil; Dexmedetomidine; Propofol; Bupivacaine; Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol-dexmedetomidine (Other): Propofol-dexmedetomidine Bupivacaine; Lidocaine (local anaesthetics) Epinephrine (with local anaesthetics for skin infiltration)
  Interventions: Drug: Dexmedetomidine; Drug: Propofol; Drug: Bupivacaine; Drug: Lidocaine; Drug: Epinephrine
- Propofol-remifentanil (Other): Propofol-remifentanil Bupivacaine; Lidocaine Epinephrine (with local anaesthetics for skin infiltration)
  Interventions: Drug: Remifentanil; Drug: Propofol; Drug: Bupivacaine; Drug: Lidocaine; Drug: Epinephrine

INTERVENTIONS:
Drug: Remifentanil — Remifentanil used for conscious sedation.
  Arms: Propofol-remifentanil
Drug: Dexmedetomidine — Dexmedetomidine used for conscious sedation.
  Arms: Propofol-dexmedetomidine
Drug: Propofol — Used for conscious sedation.
Drug: Bupivacaine — Local anaesthetics
Drug: Lidocaine — Local anaesthetic
Drug: Epinephrine — With local anaesthetic for skin infiltration.

SUMMARY:
Sixty patients were randomly allocated into two groups, group PD and group PR, thirty patients in each group. Patients in PD group received propofol and dexmedetomidine intravenous infusion and patients in PR group received propofol and remifentanil intravenous infusion. Sedation score and patients' satisfaction, surgeon satisfaction, heart rate, mean arterial blood pressure, oxygen saturation, and side effects such as respiratory depression, nausea, vomiting, airway obstruction, and oxygen desaturation were recorded.

DETAILED DESCRIPTION:
After approval from the ethics committee of Menoufia University Hospitals and informed written consent, the present study was conducted on sixty patients of both sexes. Patients' age was between 18-50 years, American society of anesthesiologists (ASA) I and II and scheduled for awake craniotomy for treatment of epilepsy. Exclusion criteria included patients with history of allergy to any of the drugs used for the study, patients with alcohol or substance abuse, pregnant females, patients with mental instability, morbid obese patients, and patients with liver, kidney, or cardiac comorbidities.

Patients were randomly allocated using computerized software into two groups, thirty patients in each group to receive intra-operative either propofol-dexmedetomidine (PD group) or propofol-remifentanil (PR group) intravenous infusion. All patients received their routine treatment for epilepsy at their scheduled time before surgery. All patients were fully monitored intra-operatively for heart rate, non-invasive blood pressure, oxygen saturation, respiratory rate, and bi-spectral index (BIS). Oxygen was supplied to all patients via nasal cannula peri-operatively.

Anaesthesia was achieved by regional scalp block and IV sedation. Regional blockade of the scalp was performed using bupivacaine 0.5% and 2% lidocaine with epinephrine 1/200.000. The branches of the cranial nerves blocked were supratrochlear, supraorbital, auriculotemporal, greater and lesser occipital, great auricular, zygomatic, and infraorbital nerves. Supplemental local anesthetic solution was used to infiltrate along the incision lines prior to skin incision. During craniotomy, a mixture of 0.25% bupivacaine and lidocaine1% without epinephrine was used to anesthetize the dura mater. The maximum dose of lidocaine used did not exceed 4.5 mg kg -1 and for bupivacaine 3 mg kg -1.

All patients received propofol 1% with a starting intravenous infusion dose of 250 μg kg-1 min-1 for 15 min and then basal infusion dose at 50 μg kg-1min-1. Sedation was achieved for group PD by a combination of propofol and dexmedetomidine with a starting infusion dose of 1ug kg-1 hr -1 for 15 min, and then titrated down to 0.2μ g kg-1 hr-1.

In PR group, IV sedation was achieved by a combination of propofol and remifentanil at an initial bolus dose of 0.5 μg.kg-1 over 60 seconds and then a basal infusion of 0.1μg kg-1 min1. Insufficient sedation in both groups was treated with boluses of 250 μg kg-1 propofol. The total amount of propofol used in both groups was recorded.

Sedation was assessed using Ramsay sedation score.6 Patient scored (1) if was anxious, agitated, or restless. Patient scored (2) if was cooperative, oriented and tranquil. Score 3 was for patients responded to command only. Score (4) for patients exhibited brisk respond to light glabellar tap or loud auditory stimulus. Score (5) for patients exhibited a sluggish response to light glabellar tap or loud auditory stimulus. Score (6) was for patients exhibited no response. Score (1) means inadequate sedation, score (2 to 4) means acceptable sedation, and score (5) or (6) means excessive sedation. Bi-spectral index (BIS) was connected to all patients and recorded every half an hour intra-operatively until the end surgery.

For intraoperative neurophysiologic monitoring propofol infusion was stopped for 15 minutes to avoid interference.

Side effects such as respiratory depression (respiratory rate less than 8/min), nausea, vomiting, airway obstruction, oxygen desaturation (oxygen saturation less than 90 %), and hypotension or hypertension (20% decrease or increase from the base line) were recorded. In case of apnea, respiratory depression, oxygen desaturation, and airway obstruction or hypotension all infusions were stopped until normalization and then the infusion resumed at half the basal rate. Vomiting was treated with 4mg intravenous ondansetron and the total ondansetron consumption was recorded for both groups.

If intraoperative convulsions occurred at any time IV thiopental sodium was given at a dose 1-2 mg kg-1. General anaesthesia was given if indicated and the patient was removed from the study. The excluded patients were replaced according to the schedule of randomization to keep the number of the two groups. Indications for general anesthesia were failure of the regional block, marked patient irritability, severe airway obstruction required intubation, uncontrolled convulsions, and haemodynamic instability.

Patient's satisfaction was recorded using a score ranging from 0 not satisfied and 10 totally satisfied. Surgeon satisfaction regarding the operative conditions and the anesthetic technique was recorded as 0 very bad operative conditions, 1 moderate, and 2 good.

Statistical analysis Sample size calculation was calculated using graphed instant statistics version 3. Based on previous research, dexmedetomidine was expected to produce a decrease in the heart rate by about 10 beats /minute with a standard deviation of 10 and by choosing 5% level of significance and power of 90% the calculated sample size was 22 so that, the sample size used in the study was 30 patients to ensure reliable results.

Data were analyzed using SPSS 19 program. Student t-test was used for comparing data between the two groups. Chi square test was used to compare the incidence of side effects. P value of less than 0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients require conscious sedation for epilepsy surgery

Exclusion Criteria:

* Patients refusal, allergy to drugs used, and uncooperative patients.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were excluded if they refused to be included in the study.
Period: Overall Study
Arm/Group | Propofol-dexmedetomidine | Propofol-remifentanil
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol-dexmedetomidine | Propofol-remifentanil | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (10.5) | 33.4 (10.5) | 33 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 17 | 16 | 33
Region of Enrollment [Number; unit: participants]
  Egypt | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Patients Satisfaction
Description: Patient's satisfaction was recorded using a score ranging from 0 for not satisfied to 10 for totally satisfied.
Time Frame: 1 hour after the operation
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Conscious sedation1: Propofol-dexmedetomidine Bupivacaine; Lidocaine (local anaesthetics) Epinephrine (with local anaesthetics for skin infiltration)
  Dexmedetomidine: Dexmedetomidine used for conscious sedation.
  Propofol: Used for conscious sedation.
  Bupivacaine: Local anaesthetics
  Lidocaine: Local anaesthetic
  Epinephrine: With local anaesthetic for skin infiltration.
- Conscious sedation2: propofol-remifentanil Bupivacaine; Lidocaine Epinephrine (with local anaesthetics for skin infiltration)
  Remifentanil: Remifentanil used for conscious sedation.
  Propofol: Used for conscious sedation.
  Bupivacaine: Local anaesthetics
  Lidocaine: Local anaesthetic
  Epinephrine: With local anaesthetic for skin infiltration.
Arm/Group | Conscious sedation1 | Conscious sedation2
Number analyzed (Participants) | 30 | 30
score on a scale | 6.33 (1.36) | 6.45 (1.41)

ADVERSE EVENTS:
Time Frame: During the operation, on average 3 hours.
Description: Apnea and airway obstruction.
Arm/Group | Propofol-dexmedetomidine | Propofol-remifentanil
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes